CLINICAL TRIAL: NCT06837675
Title: Effect of High Tone Power Therapy on Bladder Disturbance in Patients With Multiple Sclerosis
Brief Title: Effect of High Tone Power Therapy on Bladder Disturbance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Hussien Samy, physical therapist, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REC/012/005399
Record Dates: First submitted 2025-01-25; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: overactive bladder
MeSH Terms: conditions — Multiple Sclerosis; Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group 1 (Experimental): twenty patients will receive High tone power therapy and selected physical therapy program 36 sessions 3 times per week for 3 months.
  Interventions: Device: high tone power therapy; Other: selected physical therapy program
- Control group 2 (Active Comparator): twenty patients will receive a selected physical therapy program only 36 sessions 3 times per week for 3 months.
  Interventions: Other: selected physical therapy program

INTERVENTIONS:
Device: high tone power therapy — High tone Power therapy (HiToP191-H) device is a new electrotherapy technology. Its primary impact on the body is to provide energy to the body to activate cells and rebuild it. It can cause an oscillation or vibration that promotes metabolism, nand erve regeneration and relieves pain by dispersing pain and inflammation mediators, nutrients, and waste products
  Arms: Study group 1
Other: selected physical therapy program — selected physical therapy protocol for 45 minutes 3 times per week for 3 months in form of pelvic floor exercises and core stability exercise

SUMMARY:
This study is conducted to investigate the effect of high-tone power therapy on improving bladder function and quality of life in patients with MS.

DETAILED DESCRIPTION:
Inflammation, demyelination, gliosis, and neuronal loss are all components of multiple sclerosis (MS), is a chronic autoimmune disease that affects the central nervous system (CNS). Myelinated axons in the CNS are the target of MS attacks, which can cause varying degrees of damage to both myelin and axons ). MS affects 2.3 million people worldwide. MS is often diagnosed between the ages of 20 and 50 years, with females experiencing it more often than males. Among the most common MS symptoms are disorders of motor function and gait, spasticity, and sensory challenges including visual problems

. which are causes of disability that are possible to identify by observing from the outside. However, other frequent and disabling symptoms are invisible, including fatigue, cognitive deficits and decline, emotional distress, and pain. Dysfunction of the bladder and bowel are also hidden consequences of MS but rank among the most frequent and troublesome symptoms. it is estimated that 75-90 % of MS will experience bladder problems and up to 50 % of MS will experience bowel problems at some stage in their life. Bladder dysfunction is reported to cause major limitations in one's daily life, and contribute to decreased satisfaction with one's life situation and health Lesions above the pontine micturition center are usually associated with neurogenic detrusor overactivity (NDO), characterized by involuntary detrusor contractions 3 (urgency, frequency, urge incontinence, and no or low post-void residual urine).

Urgency is the sudden desire and intense sensation of needing to pass urine; frequency is the need to urinate many times during the day or at night (nocturia) or both, but in normal or less-than-normal volumes; urge incontinence is an involuntary urine leak while having symptoms of urgency. High-tone power therapy (HTT) is a unique characteristic of electrotherapy. It uses intermediate frequency, metal-compatible alternating current whose frequency oscillates between approximately 4000 Hz and 33000 Hz and intensity is adjusted, unlike traditional electrotherapies such as TENS. Its main effects are introducing energy into the body to activate cells, producing an oscillation or vibration in the cells and tissues to promote metabolism, normalizing the cell metabolism and nerve regeneration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with MS complaining of bladder disturbance referred by neurologist with a urodynamic study 2. Patients age will be ranged from 20 to 50 years old 3. Body mass index from (18.5 to 24.9) 4. Score of disability 2 to 6 according to EDSS 5. Patients with overactive bladder at least 6 months before the study 6. The severity of overactive bladder OAB will range from 6 to 10 according to overactive bladder symptom score (moderate stage) (OABSS). 7. All the patients will be in the remission period. 8. All the patients will receive the same medical treatment. 9. All the drugs that interfere with bladder function will be stopped. 10. Patients must be medically stable. 11. Patients able to respond to verbal instructions

Exclusion Criteria:

* 1. Unstable cardiac condition (MI, severe cardiac failure) 2. Systemic diseases (DM, RA, AKI) 3. Patients with musculoskeletal deformities 4. Any tumor affects the lumber spine 5. Patients with cognitive problems 16 6. Open wound, burn, and loss of sensation 7. Patients with metal implants 8. Any other diseases that may cause OAB, such as inflammatory or urinary tract infections, Prostatitis in male or Female genital disorders 9. Patients with a history of abdominal or bladder surgeries or diseases 10. MS patients in acute relapse stage 11. Patients with diabetic polyneuropathy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
over active bladder symptom score (OABSS) | the test will be done 3 days before the beginning of the study and 3 days after completion of the study.
  Assessment scale for overactive bladder syndrome. It consists of 4 questions about frequency, nocturnal, urgency, and urge incontinence. Total score from 0 to 15
Urodynamic study | the test will be done 3 days before the beginning of the study and 3 days after completion of the study.
  The urodynamic study is the golden objective for assessing the bladder's physiological and pathological functions. The test involves an invasive assessments of bladder storage function and bladder emptying function
MS bladder check tool | the test will be done 3 days before the beginning of the study and 3 days after completion of the study.
  it is a check tool that aims to improve the management of people with Multiple sclerosis.
The international Consultation on Incontinence Questionnaire Short Form (ICIQ-UI) | the test will be done 3 days before the beginning of the study and 3 days after completion of the study.
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided